CLINICAL TRIAL: NCT06784466
Title: Coherent Sine Burst Electroporation (CSE) Ablation System US Investigational Device Exemption (IDE) Study for Patients With Atrial Fibrillation
Brief Title: Coherent Sine Burst Electroporation (CSE) Ablation System US IDE Study for Patients With Atrial Fibrillation
Acronym: COHERENT-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arga Medtech SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Persistant Atrial Fibrillation; Paroxysmal AF
Keywords: atrial fibrillation; ablation; coherent sine-burst; electroporation; pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Non-randomized, multi-center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Paroxysmal AF (Experimental): Patients with paroxysmal AF will receive treatment using the Arga Medtech Coherent Sine-Burst Electroporation ablation system to achieve pulmonary vein isolation.
  Interventions: Device: Argá Medtech Coherent Sine-Burst Electroporation (CSE) Ablation System
- Persistent AF (Experimental): Patients with persistent AF will receive treatment using the Arga Medtech Coherent Sine-Burst Electroporation ablation system to achieve pulmonary vein isolation.
  Interventions: Device: Argá Medtech Coherent Sine-Burst Electroporation (CSE) Ablation System

INTERVENTIONS:
Device: Argá Medtech Coherent Sine-Burst Electroporation (CSE) Ablation System — Ablation using the Argá Medtech Coherent Sine-Burst Electroporation (CSE) Ablation System

SUMMARY:
To evaluate the safety and effectiveness of the Argá Medtech CSE Ablation System in the treatment of atrial fibrillation.

DETAILED DESCRIPTION:
A prospective, multi-center, non-randomized, unblinded pre-market study designed to provide clinical data to support regulatory approval of the Argá Medtech CSE Ablation System for the ablation of atrial fibrillation and adjunctive use for additional atrial ablation. Patients with a history of drug refractory, recurrent, symptomatic, paroxysmal atrial fibrillation (PAF) or persistent atrial fibrillation (PersAF) will, at a minimum, undergo ablative intervention of the pulmonary veins.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 and 80 years, or older than 18 if required by local law.
2. Diagnosis of drug refractory, recurrent, paroxysmal or persistent AF:

   a. Symptomatic paroxysmal AF that is less than 7 days in continuous duration, documented by the following: i. Physician documentation of symptomatic recurrent PAF (2 or more episodes) within 6 months prior to enrollment AND ii. At least 1 documented AF episode from any form of rhythm monitoring within 12 months prior to enrollment.

   b. Symptomatic persistent AF that is sustained beyond 7 days and less than 1 year (≥ 7 and ≤ 365 days), documented by the following: i. Physician documentation of at least 1 symptomatic persistent AF episode within 6 months prior to enrollment.

   ii. Either a 24-hour continuous ECG recording documenting continuous AF OR 2 ECGs from any regulatory cleared rhythm monitoring device showing continuous AF taken at least 7 days apart, within 6 months prior to enrollment.
3. Effectiveness failure of, intolerance to, or a specific contraindication to at least one Class I or III anti-arrhythmic drug.
4. Willing and able to give informed consent.
5. Willingness, ability, and commitment to participate in baseline, follow-up, and rhythm monitoring evaluations for the full length of the study.
6. Life expectancy >1 year.

Exclusion Criteria:

1. In the opinion of the Investigator, any known contraindication to an AF ablation (including present left atrial [LA] thrombus), trans-esophageal echocardiogram (TEE) or computed tomography (CT) scan, or anticoagulation.
2. Any duration of continuous AF lasting longer than 12 months.
3. History of any previous left atrial ablation or surgical procedure, including prior left atrial appendage closure.
4. AF secondary to electrolyte imbalance, thyroid disease, alcohol, or any other reversible or non-cardiac cause.
5. Left ventricular ejection fraction (LVEF) < 35% within 6 months of enrollment (e.g. transthoracic echocardiogram (TTE), multiple-gated acquisition (MUGA), magnetic resonance imaging (MRI), nuclear stress test).
6. New York Heart Association (NYHA) Class III or IV.
7. Left atrial diameter > 5.0 cm (anteroposterior) within 6 months of enrollment (MRI, CT, TTE, TEE, or physician's note) or non-indexed volume >100mL if left atrial diameter is not available.
8. Current or anticipated implant of a permanent pacemaker, implantable cardioverter or resynchronization device, interatrial baffle, foramen ovale occluder, LA appendage closure, or active implantable/insertable cardiac loop recorder/monitor at the time of the ablation procedure.
9. Body mass index (BMI) >40.
10. Patients who have not been on anticoagulation therapy for at least 3 weeks prior to the Index Procedure.
11. Previous cardiac surgery, myocardial infarction, percutaneous coronary intervention or angioplasty (PCI/PTCA) or coronary artery stenting within 3 months prior to enrollment.
12. Symptomatic valvular disease, history of cardiac valve surgery, or prosthetic mitral and tricuspid valve(s).
13. Presence of pulmonary vein abnormalities of stenosis or stenting.
14. Primary pulmonary hypertension.
15. Uncontrolled or untreated hypertension (two measurements of >180mmHg systolic or >110 mmHg diastolic at baseline).
16. Pre-existing hemi-diaphragmatic paralysis.
17. Renal insufficiency with an estimated glomerular filtration rate (eGFR) < 40 mL/min/1.73 m2, or any history of renal dialysis or renal transplant.
18. Rheumatic heart disease.
19. Unstable angina or ongoing myocardial ischemia.
20. Hypertrophic cardiomyopathy, advanced restrictive cardiomyopathy, or severe left ventricular hypertrophy (left ventricular thickness >15mm).
21. History of blood clotting or bleeding disease (e.g., thrombocytosis).
22. History of documented cerebral infarction, transient ischemic attack, or systemic embolism within 6 months prior to enrollment.
23. Active systemic infection.
24. Active malignancy or history of treated malignancy within 12 months of enrollment (other than cutaneous basal cell or squamous cell carcinoma, or non-metastatic prostate or breast cancer with life expectancy remaining >1 year).
25. Pregnant or lactating (current or anticipated during study follow-up).
26. Current enrollment in any other clinical study where testing or results from that study may interfere with the procedure or outcomes measurement for this study.
27. Any other condition that, in the judgment of the Investigator, makes the patient:

    1. Unlikely to benefit from an AF ablation procedure (e.g., advanced infiltrative cardiomyopathies, severe mitral stenosis or regurgitation, and/or cor pulmonale, etc.), or
    2. A poor candidate for the study (e.g., vulnerable patient population, mental illness, addictive disease, terminal illness, and extensive travel away from the research center).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of Participants With at Least One Primary Safety Event. | Up to 180 days
  Primary safety events are:
  Within 7 days of the index procedure:
  * Complete heart block
  * Coronary spasm
  * Myocardial infarction
  * Peripheral or organ thromboembolism
  * Stroke
  * Transient ischemic attack
  * Unresolved phrenic nerve palsy
  * Vascular access complications
  * Pericarditis
  Within 30 days of the index procedure:
  * Acute renal failure
  * Cardiac tamponade / perforation
  * Cardiovascular or pulmonary Pulsed Field Ablation (PFA)-related hospitalization
  * Death
  * Gastroparesis
  * Major bleeding
  Within180 days of the index procedure:
  * Pulmonary vein stenosis (≥70% diameter reduction)
  * Esophageal perforating complications
Effectiveness: Number of Participants With Treatment Success. | Up to 12 months
  Treatment success is defined as freedom from treatment failure.
  1. Acute Procedural Success and
  2. Chronic Success:
     * Documented atrial fibrillation (AF), atrial flutter (AFL), or atrial tachycardia (AT) on a 12-lead electrocardiogram (ECG), event monitor, or Holter monitor after the 90-day Blanking Period
     * Re-ablation in the left atrium for AF, AFL, or AT
     * Any electrical cardioversion for AF, AFL, or AT
     * Any Class I or III antiarrhythmic (AAD) dose increase from the historic maximum ineffective dose prior to the Index Procedure or initiation of any new Class I or III AAD.

SECONDARY OUTCOMES:
Quality of Life - Change in EQ-5D-3L Score | Baseline to 12 months post-ablation
  Change in EQ-5D-3L score (12-month score - baseline score). The Euroqol EQ-5D-3L questionnaire (3L version) is a standardized instrument for measuring general health status. The Euroqol EQ-5D-3L questionnaire (which consists of a 5-question survey and a visual analog scale) has a composite score based on the 5-question survey that ranges from 0 (least healthy) to 1 (most healthy).
Quality of Life - Change in The AF Effect on Quality-of-Life questionnaire (AFEQT) Score | Baseline to 12 months post-ablation
  Change in AFEQT score (12-month score - baseline score). The AFEQT questionnaire is an atrial fibrillation (AF) specific health-related quality of life questionnaire to assess the impact of AF on a subject's life. The overall score ranges from 0 - 100, with 0 corresponding to complete disability and 100 corresponding to no disability.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (15):
  - Grandview, Birmingham, Alabama
  - Banner University Med Ctr, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - UCSD, San Diego, California
  - Ascension / St. Vincent's Jacksonville, Jacksonville, Florida
  - Emory, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Kansas City Heart Rhythm Institute (KCHRI), Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - TriHealth Cincinnati, Cincinnati, Ohio
  - Trident Medical Center, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Methodist, San Antonio, Texas
- Belgium (2):
  - AZorg Aalst, Aalst
  - Jessa Ziekenhuis, Hasselt
- Croatia (2):
  - KBC Split, Split
  - KBC Zagreb, Zagreb
- Czechia (3):
  - Neuron Medical s.r.o., Brno, Czech Republic
  - Institut klinické a experimentální medicíny (IKEM), Prague, Czech Republic
  - Nemocnice Na Homolce, Prague
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No
data will be published in aggregate